CLINICAL TRIAL: NCT02724332
Title: A Randomized Controlled Study on the Effect of Adjuvant Anti-recurrence Treatment With Rapamycin on Early-stage HCC With Overexpression of ASPH After Radical Surgery.
Brief Title: Adjuvant Anti-Recurrence Treatment With Rapamycin on Early-stage HCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZD201206003-P1
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Rapamycin
Keywords: Aspartate beta hydroxylase; transcatheter arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): Patients will be treated with radical hepatectomy only.
- transcatheter arterial chemoembolization (Active Comparator): Patients will be treated with TACE
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — 2mg,po,bid
  Arms: transcatheter arterial chemoembolization

SUMMARY:
To evaluate the clinical effect of rapamycin combined with TACE on early-stage HCC with overexpression of ASPH after radical surgery using randomized controlled study and provide a new anti-recurrence treatment for HCC patients after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Via clinical diagnosis and confirm it is primary liver cancer
2. Pathological evidence of HCC
3. Estimate tumor can gain treatment of curing operation
4. No evidence for extrahepatic metestasis
5. liver function ：Child-Pugh A/B
6. BCLC stage：0/1；TNM stage：Ⅰ

Exclusion Criteria:

1. reject to attend；
2. impossible to come to our hospital for physical examination regularly.
3. cancer epitome、seed focus、lymph node or distant metastasis
4. Blood clotting function hindrance; 5, Patients with other diseases which may affect the treatment mentioned.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years

SECONDARY OUTCOMES:
Time to recurrence | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China